CLINICAL TRIAL: NCT04390958
Title: Phase II Study of Neoadjuvant Chemotherapy With Nab-paclitaxel Plus Cisplatin and Capecitabine for Locally Advanced Thoracic Esophageal Squamous Cell Carcinoma
Brief Title: Neoadjuvant Chemotherapy With Nab-paclitaxel Plus Cisplatin and Capecitabine for Locally Advanced Thoracic Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Aiping Zhou, Vice director of Department of Medical Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC-003475
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — 130-nm albumin-bound paclitaxel; Cisplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant chemotherapy group (Experimental): Total 6 perioperative chemotherapy composed of nab-paclitaxel, cisplatin and capecitabine every 21 days
  Interventions: Drug: nab-paclitaxel; Drug: Cisplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: nab-paclitaxel — 125mg/m2 ivgtt d1、d8
Drug: Cisplatin — 60mg/m2 ivgtt d1 or d1-2
Drug: Capecitabine — 1750mg/m2 po bid d1-14

SUMMARY:
Surgical resection is currently the major treatment for esophageal carcinoma while disease progression still occurred in most cases within 3 years. The rate of local recurrence and distant metastases could reach nearly 40% to 60%. The neoadjuvant chemotherapy could significantly improve resection rate and overall survival after surgery. Squamous cell carcinoma is the most common histology in Asia. JCOG9907 trial performed in Japan confirmed that compared to surgery plus adjuvant chemotherapy, the combination of neoadjuvant chemotherapy and surgery could further prolong overall survival. The regimen of cisplatin and fluorouracil is a classic effective option in combination therapy for esophageal carcinoma. Nanoparticle albumin-bound (nab)-paclitaxel is a novel taxane and has better efficacy in esophageal carcinoma treatment. We try to evaluate the efficacy and safety of neoadjuvant chemotherapy with nab-paclitaxel plus cisplatin and capecitabine for locally advanced thoracic esophageal squamous cell carcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologic pathological or cytological diagnosis of squamous cell carcinoma of esophagus
* Age ranges from 18 to 70 years
* Patients must not have received any prior anticancer therapy
* Preoperative stage cT2N+M0, cT3-4aN0/N+M0 thoracic esophageal squamous cell carcinoma evaluated by MDT consultation based on imaging examinations
* Eastern cooperative oncology group (ECOG) performance status of 0 to 1
* Signed informed consent document on file
* Females with childbearing potential must have a negative serum pregnancy
* Adequate organ function to receive esophagectomy including the following:

Bone marrow: absolute white blood cells count ≥3.0×10^9/L, absolute neutrophil count (ANC) ≥1.5×10^9/L, platelets ≥100×10^9/L, haemoglobin ≥90g/L; Hepatic: total bilirubin ≤1.5 times upper limit of normal (ULN), alanine transaminase (ALT) and aspartate transaminase (AST) ≤2.5 times ULN; Renal: calculated creatinine clearance rate≥80ml/min

* For childbearing potential males and females, who have agreed with contraception from start of investigational drug administration to 6 months after last dose of investigational drug
* Patients who have no contraindication of nab-paclitaxel, cisplatin or capecitabine

Exclusion Criteria:

* Patients who may develop tracheoesophageal fistula or aortoesophageal fistula
* Patients who have received allogeneic organ or stem cell transplants
* Patients with uncontrolled diabetes mellitus, any serious or unstable medical condition or mental illness
* Patients with preexisting or a history of ≥ Grade II peripheral neuropathy
* Pregnant or breast feeding
* Patients who take part in clinical trials of other drugs or biological therapy within 4 weeks before enrollment
* Prior invasive malignancy in 5 years (except for curable carcinoma in situ of cervix and non-melanoma skin cancer)
* Patients with digestive tract obstruction or metabolic dysfunction which may influence oral absorption of capecitabine
* Patients with supraclavicular lymph node metastasis, celiac lymph node metastasis except for pericardial and left gastric lymph node metastasis
* Patients with evidence of distant metastases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | 2 year
  No cancer cells in primary tumor and all lymph nodes resected are observed by pathologists

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 2 year
  Objective response rate is defined as the rate of patients with at least a 30% decrease in the sum of the LD (longest diameter) of target lesions, which include complete response (CR) or partial response (PR)
R0 resection rate | 2 year
  The ratio of the patients with surgical R0 resection over the of patients who receive surgery
Major Pathological Response (MPR) rate | 2 year
  MPR is defined as 10% or fewer viable cancer cells in the hematoxylin and eosin (H&E)-stained slides from the resected tumor following neoadjuvant treatment
Overall survival (OS) | From date of enrollment until the date of death from any cause, assessed up to 24 months
  Time from enrollment to death
Disease free survival (DFS) | From date of enrollment until the date of death or recurrence, assessed up to 24 months
  From the day of surgery with R0 resection to recurrence or death of any reasons
Progression-free survival (PFS) | From date of enrolment until the date of first documented disease progression or date of death from any cause, whichever came first, assessed up to 24 months
  number of participant with disease progression
Recurrence rate | 2 year
  number of participant with disease recurrence
Treatment-emergent adverse events | 2 year
  From the day of neoadjuvant therapy to 30 days after surgery or within 90 days after last neoadjuvant treatment. To evaluate the incidence of TEAE, rate of grade 3 and 4 TEAE (CTCAE 5.0), rate of surgery delay over 30 days and/or inoperable patients
Surgical complications | Within the first 90 days after the start of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Shugeng Gao, MD, Principal Investigator — Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

REFERENCES:
- [Derived] Zhang W, Chen X, Xue L, Jiang Z, Qu D, Yang Z, Qin J, Wang Z, Zhang M, Li Y, Zhou A, Gao S. Neoadjuvant chemotherapy with albumin-bound paclitaxel plus cisplatin and capecitabine for locally advanced esophageal squamous cell carcinoma: a phase 2 clinical trial. Int J Surg. 2025 Jun 1;111(6):3831-3837. doi: 10.1097/JS9.0000000000002375. Epub 2025 May 12. PMID 40358628